CLINICAL TRIAL: NCT06364397
Title: Efficacy of ERCP in the Diagnosis and Treatment of Idiopathic Recurrent Acute Pancreatitis: a Randomized Controlled Trial
Brief Title: Efficacy of ERCP in the Diagnosis and Treatment of Idiopathic Recurrent Acute Pancreatitis
Acronym: ESPRIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Collaborators: Peking Union Medical College Hospital (Other); First People's Hospital of Hangzhou (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Professor, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ESPRIT202403
Record Dates: First submitted 2024-04-03; First posted 2024-04-15 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Recurrent Acute Pancreatitis
Keywords: Recurrent acute pancreatitis; Idiopathic; ERCP; Sphincterotomy
MeSH Terms: conditions — Pancreatitis | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERCP group (Experimental): Participants will undergo ERCP. Indomethacin will be administered rectally before procedure in participants with no known allergy to indomethacin. If the etiology of the participant is clearly defined during ERCP, the corresponding endoscopic treatment procedure will be performed. For others whose etiology are still unclear, pancreatic sphincterotomy and small caliber prophylactic pancreatic duct stent replacement will be performed. The participants will be observed closely after ERCP and record complications. Abdominal X-rays will be taken 2 weeks after ERCP to confirm spontaneous passage of the pancreatic duct stent, and the stent will be removed via gastroscopy if it still in place. Participants will accept health education and conservative management of clinical routines. Follow-up visits for participants occurred at 3, 6, 9 and 12 months after enrollment.
  Interventions: Procedure: ERCP; Combination Product: Health education and conservative management of clinical routines
- conservative treatment group (Active Comparator): Participants will be given health education and conservative management of clinical routines. Follow-up visits for participants occurred at 3, 6, 9 and 12 months after enrollment.
  Interventions: Combination Product: Health education and conservative management of clinical routines

INTERVENTIONS:
Procedure: ERCP — Participants will undergo ERCP and indomethacin will be administered rectally before procedure in participants with no known allergy to indomethacin. If the etiology of the participant is clearly defined during ERCP, the corresponding endoscopic treatment procedure will be performed. For others whose etiology are still unclear, pancreatic sphincterotomy and small caliber prophylactic pancreatic duct stent replacement will be performed. The participants will be observed closely after ERCP and record complications. Abdominal X-rays will be taken 2 weeks after ERCP to confirm spontaneous passage of the pancreatic duct stent, and the stent will be removed via gastroscopy if it still in place.
  Arms: ERCP group
Combination Product: Health education and conservative management of clinical routines — Participants will be given health education and conservative management of clinical routines. Clinical management is based on the pancreatic endocrine and exocrine function.

SUMMARY:
The goal of this clinical trial is to learn if endoscopic retrograde cholangiopancreatography (ERCP) works to treat idiopathic recurrent pancreatitis (IRAP) in adults. It also clarify the efficacy of ERCP in the diagnosis of IRAP. The main questions it aims to answer are:

Does ERCP reduce the frequency of pancreatitis episodes in IRAP patients? Does ERCP contribute to identify the etiology of IRAP patients?

Participants will be randomly allocated to receive ERCP (pancreatic sphincterotomy and pancreatic stent placement) or conservative treatment and be followed for 1 year.

DETAILED DESCRIPTION:
Recurrent acute pancreatitis (RAP) is defined as 2 or more distinct episodes of acute pancreatitis (AP) with complete resolution between each episode, and absence of irreversible structural and functional changes in pancreas. RAP has an estimated annual incidence of 8-10 per 100,000 and the recurrence rate is as high as 10-30% in AP patients. At present, biliary, alcoholic and hypertriglyceridemia are common causes of RAP. There are also a variety of causes that may contribute to recurrent episodes of AP, such as gene mutations, pancreas divisum, ampullary neoplasms and sphincter of Oddi dysfunction. About 80% of RAP patients can be identified through routine clinical investigations (include proper history, physical examination, imaging examination); however, the etiology in up to 20% of cases still not be clarified and these patients is called idiopathic recurrent acute pancreatitis (IRAP).

Endoscopic retrograde cholangiopancreatography (ERCP) is an important minimally invasive treatment for pancreatic diseases. However, the role of ERCP in IRAP patients with normal biliary and pancreatic anatomy remains controversial and there is a lack of high-quality clinical research evidence on endoscopic treatment of IRAP. In a small sample size (N=34) open-label randomized controlled study, IRAP patients were assigned to the experimental group with pancreatic duct stent placement and the control group with selective pancreatograms but no stent. This study demonstrated that stent placement was able to reduce the recurrence rate of AP (53% vs 11%, P < 0.02). Coté et al performed an open-label randomized trial (N=89) of ERCP with sphincter of Oddi manometry for IRAP patients. Among patients with pancreatic sphincter dysfunction, they found that biliary sphincterotomy and combination of biliary and pancreatic sphincterotomy have similar effects in preventing recurrence of AP, and there was also no significant difference between biliary sphincterotomy and sham surgery in patients with normal sphincter of Oddi manometry. However, some retrospective studies had shown that sphincterotomy works to reduce the recurrence rate of acute pancreatitis.

Currently, there is a shortage of high-quality evidence, and the wide variation in different study designs has led to controversial conclusions. Given the long-standing controversy, we propose to conduct a randomized controlled trial to investigate the efficacy of ERCP in the diagnosis and treatment of Idiopathic recurrent acute pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 70 years.
2. Patients diagnosed with IRAP:

   1. Previously experienced 2 or more distinct episodes of acute pancreatitis (AP) with complete resolution between each episode, and absence of irreversible structural and functional changes in pancreas. The diagnosis of AP is based on the Atlanta criteria and is documented in the medical record.
   2. The etiology of RAP remains undetermined after routine clinical investigations, including history, laboratory examination, imaging examination (CT, MRI/MRCP, EUS). Patients who still have AP episodes after elimination of the etiology also be included.
3. At least 1 episode of AP one year prior to enrollment.
4. Consent to participate in the study and sign the informed consent form.

Exclusion Criteria:

1. Prior sphincter intervention.
2. Not recovered from prior AP attack.
3. Prior pancreatic surgery.
4. Contraindications to ERCP.
5. Major mental illness or serious health problems that are not suitable for participation in the study.
6. Pregnancy or plan for pregnancy within 12 months of enrollment.
7. Other conditions that inappropriate to participant in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate of AP | 1 year after enrollment
  Proportion of patients with at least one episode of AP 1 year after enrollment (AP within 1 month of the index ERCP was excluded).

SECONDARY OUTCOMES:
Ratio of reduced AP episodes | 1 year after enrollment
  Ratio of the reduced AP episodes (1 year before and after enrollment) to the AP episodes in 1 year before enrollment. AP within 1 month of the index ERCP was excluded.
Proportion of patients with reduced AP episodes | 1 year after enrollment
  Proportion of patients whose AP episodes reduced (1 year before and after enrollment). AP within 1 month of the index ERCP was excluded.
Severity of AP | 1 year after enrollment
  Proportion of patients with different severity of AP that according to the Atlanta criteria.
Evaluation of quality of life | 1 year after enrollment
  Evaluate by the Medical Outcomes Study 36-Item Short Form Health Survey (SF-36) that measures health on eight dimensions. For each dimension, item scores are coded, summed, and transformed into a scale from 0 (worst health) to 100 (best health).
Evaluation of psychological condition | 1 year after enrollment
  Evaluate by the Depression Anxiety Stress Scale (DASS-21), which consists of 21 items with a total score of 0-63. The higher the score, the more serious the adverse psychological state of the patient.
Proportion of patients diagnosed by ERCP. | 1 year after enrollment
  Proportion of patients whose etiology was identified by ERCP.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoshen Li, M.D., Study Chair — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guda NM, Trikudanathan G, Freeman ML. Idiopathic recurrent acute pancreatitis. Lancet Gastroenterol Hepatol. 2018 Oct;3(10):720-728. doi: 10.1016/S2468-1253(18)30211-5. PMID 30215363
- [Background] Machicado JD, Yadav D. Epidemiology of Recurrent Acute and Chronic Pancreatitis: Similarities and Differences. Dig Dis Sci. 2017 Jul;62(7):1683-1691. doi: 10.1007/s10620-017-4510-5. Epub 2017 Mar 9. PMID 28281168
- [Background] Sankaran SJ, Xiao AY, Wu LM, Windsor JA, Forsmark CE, Petrov MS. Frequency of progression from acute to chronic pancreatitis and risk factors: a meta-analysis. Gastroenterology. 2015 Nov;149(6):1490-1500.e1. doi: 10.1053/j.gastro.2015.07.066. Epub 2015 Aug 20. PMID 26299411
- [Background] Ahmed Ali U, Issa Y, Hagenaars JC, Bakker OJ, van Goor H, Nieuwenhuijs VB, Bollen TL, van Ramshorst B, Witteman BJ, Brink MA, Schaapherder AF, Dejong CH, Spanier BW, Heisterkamp J, van der Harst E, van Eijck CH, Besselink MG, Gooszen HG, van Santvoort HC, Boermeester MA; Dutch Pancreatitis Study Group. Risk of Recurrent Pancreatitis and Progression to Chronic Pancreatitis After a First Episode of Acute Pancreatitis. Clin Gastroenterol Hepatol. 2016 May;14(5):738-46. doi: 10.1016/j.cgh.2015.12.040. Epub 2016 Jan 6. PMID 26772149
- [Background] Jacob L, Geenen JE, Catalano MF, Geenen DJ. Prevention of pancreatitis in patients with idiopathic recurrent pancreatitis: a prospective nonblinded randomized study using endoscopic stents. Endoscopy. 2001 Jul;33(7):559-62. doi: 10.1055/s-2001-15314. PMID 11473324
- [Background] Cote GA, Imperiale TF, Schmidt SE, Fogel E, Lehman G, McHenry L, Watkins J, Sherman S. Similar efficacies of biliary, with or without pancreatic, sphincterotomy in treatment of idiopathic recurrent acute pancreatitis. Gastroenterology. 2012 Dec;143(6):1502-1509.e1. doi: 10.1053/j.gastro.2012.09.006. Epub 2012 Sep 11. PMID 22982183
- [Background] Strand DS, Law RJ, Yang D, Elmunzer BJ. AGA Clinical Practice Update on the Endoscopic Approach to Recurrent Acute and Chronic Pancreatitis: Expert Review. Gastroenterology. 2022 Oct;163(4):1107-1114. doi: 10.1053/j.gastro.2022.07.079. Epub 2022 Aug 22. PMID 36008176
- [Background] Wehrmann T. Long-term results (>/= 10 years) of endoscopic therapy for sphincter of Oddi dysfunction in patients with acute recurrent pancreatitis. Endoscopy. 2011 Mar;43(3):202-7. doi: 10.1055/s-0030-1255922. Epub 2010 Nov 24. PMID 21108172